CLINICAL TRIAL: NCT01448083
Title: Heart/Mediastinal Ratio Study for Potential Equivalence of Heart/Mediastinal Ratios at One and Two Hours to the Traditional Heart/Mediastinal Ratio Obtained at Four Hours
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nuclear Medicine Consultants, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 11-MIBG-005
Record Dates: First submitted 2011-10-03; First posted 2011-10-07 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Neuroendocrine Tumor
Keywords: I-131 MIBG therapy; whole body I-123 MIBG scintigraphy
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neuroendocrine tumor patients
  Interventions: Other: Standard of care diagnostic MIBG scan for neuroendocrine tumor diagnosis.

INTERVENTIONS:
Other: Standard of care diagnostic MIBG scan for neuroendocrine tumor diagnosis. — Each subject will receive a 370 MBq (10 mCi ) (±10%) injection of I- 123 MIBG. Myocardial I-123 MIBG uptake will be quantitatively measured over time via planar imaging acquired at 15 minutes, one, two, four, and at 24 hours (the standard of care time point for NET patient imaging) post I-123MIBG injection.

SUMMARY:
The purpose of this study is to determine if the measurement (with a standard nuclear camera) of radioactivity normally present in the nervous system of your heart at four hours after the injection of radioactive drug for your diagnostic I-123 MIBG scan is any different than radioactivity measured in your heart at one and/or two hours after your diagnostic scan injection. If equivalent information to the conventional 4 hr H/M ratio could be collected by obtaining H/M ratios at 1 or 2 hour windows, it would greatly facilitate patient acceptance of the procedure since the requirements for obtaining a valid H/M ratio would be considerably less time-consuming.

One hour before being injected with the drug (I-123 MIBG) for your MIBG scan, you will be given a standard dose of non-radioactive iodine (Lugol's solution) to block your thyroid from receiving the small amount of radiation that is a normal part of the MIBG scan. You will then be injected with MIBG, and you will have 10 minute pictures of your chest at 15 minutes, 1 hour, 2 hours, and 4 hours in addition to the standard 24 hour pictures. These pictures will be taken in the Nuclear Medicine Section, Department of Radiology at Ochsner Medical Center-Kenner. The experimental (research) part of this study is having the extra 10-minute pictures of your chest at 15 minutes, 1 hour, 2 hours, and 4 hours. Normally, pictures are only taken 24 hours after the injection. Therefore the research is limited to the four extra pictures taken, and involve no additional injections or I-123 drug beyond that you will be receiving regardless of whether you are part of this research.

ELIGIBILITY:
Inclusion Criteria:

1. NET patients who are potential candidates for I-131 MIBG therapy, and are having whole body I-123 MIBG scintigraphy as standard of care.
2. Male or female patients ≥ 18 years of age.
3. Written informed consent from patients obtained in accordance to local guidelines.
4. History and physical exam indicating low likelihood, < 10 %, of any significant cardiac disease.
5. Echocardiogram within normal limits, including absence of valvular disease and normal LVEF.
6. Serum BNP within normal limits. -

Exclusion Criteria:

1. Patients on drugs which interfere with MIBG uptake - tricyclic antidepressants, phenylpropanolamine, pseudephredine, phenylephrine, sympathomimetics, amphetamines, reserpine, thorazine and thiothixines, calcium channel blockers, cocaine, and long-acting beta blockers.
2. >10% likelihood of any significant heart disease, including myocardial ischemia, cardiomyopathies, uncontrolled hypertension, congestive heart failure and valvular heart disease, e.g. see "Likelihood of Assessment of Coronary Artery Disease" below.
3. History of uncontrolled diabetes mellitus
4. Signs/symptoms of neurological diseases (e.g., Parkinsonian syndromes) or other disease known to affect the sympathetic nervous system.
5. Female patients who are pregnant or nursing (lactating), or adults of reproductive potential who are not using effective birth control methods. If there is any question of pregnancy, a serum bHCg will be collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuroendocrine Tumor Clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-10

PRIMARY OUTCOMES:
The heart/mediastinal ratio (H/M) at one or two hours post injection of AdreView™ (I-123 MIBG) in neuroendocrine tumor patients is equivalent to the standard 4 hr calculation. | Approximately 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Medical Center - Kenner, Kenner, Louisiana, United States